CLINICAL TRIAL: NCT00184340
Title: Secured Internet-mediated Psychotherapy With Psychiatry Patients. Software Improvement, Clinical Trials and Development of Clinical Precautions
Brief Title: Secured Internet-mediated Psychotherapy With Psychiatry Patients
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Directorate of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: FORSKPRO-ID p03000217
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Psychiatric Disorders
Keywords: eTherapy supplementary
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: eTherapy — secured e-mail system between patient and therapist
  Other Names: Treatment as usual

SUMMARY:
This is the second phase (Phase B) of the main project "Bank for Thoughts", which has the following aims:

1. Improvement of software for secured (encrypted and access-controlled) asynchronous text-based communication within health services. (Adjustments for use in psychiatry.)
2. Open clinical trials with Internet-mediated psychotherapy or counselling in out-patient child and adolescent psychiatry.
3. Development of indications and precautions for text-based Internet-mediated psychotherapy.

DETAILED DESCRIPTION:
This phase (Phase B) concentrates on qualitative evaluation of open clinical single case trials using asynchronous Internet-mediated text-dialogue for psychotherapeutic purposes.

Single patients in differing treatment phases, conditions, age and sex categories are interviewed after using Internet-contact as a supplementary tool in psychotherapy. Their therapists are interviewed as well.

The purpose is systematically gathering single-case experiences with the tool, to build a hypothesis for research and preliminary guidelines for experimental clinical use of Internet-mediated psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Motivation for e-mail contact
* Therapist evaluation for suitability

Exclusion Criteria:

* Paranoia
* Psychosis
* Eating disorders
* Addictive problems
* Denying or concealing symptoms

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Clients in CAMH services
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Rimehaug, Asst. Prof., Study Director — Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dept. of Neuroscience, Center for Child and Adolescent Mental Health
Locations (2):
- Norway (2):
  - Child Psychiatry Department, Levanger Hospital, Levanger
  - Child Psychiatry Department, St. Olav Hospital, Orkdal Site, Orkanger

REFERENCES:
- [Result] Joraas T, Rimeheug T, Birkeland MS, Arefjord K. E-therapy as a follow-up supplement to outpatient treatment of adolescents: A qualitative study of therapist experiences. Tidsskrift for Norsk Psykologforening 46(4): 355-61, 2009
- [Result] Birkeland MS, Rimehaug T, Arefjord K, Joraas T. How clients experience e-therapy as a supplement to ordinary psychotherapy. Tidsskrift for Norsk Psykologforening 46(4): 348-358, 2009.